CLINICAL TRIAL: NCT05144581
Title: Treatment of IBS in Primary Health Care: Adherence to Guidelines
Brief Title: Treatment of IBS in Primary Health Care.
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Region Örebro County (Other)
Responsible Party: Sponsor
Other Study IDs: 277071
Record Dates: First submitted 2021-11-22; First posted 2021-12-03 (Actual); Last update posted 2021-12-03 (Actual); Status verified 2021-11

CONDITIONS: Irritable Bowel Syndrome
Keywords: Irritable bowel syndrome; Functional gastrointestinal disorders
MeSH Terms: conditions — Irritable Bowel Syndrome; Gastrointestinal Diseases

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients diagnosed with IBS: Patients diagnosed with IBS within primary care in Region Örebro County 2013-2017, identified by ICD-code K.58.

SUMMARY:
The purpose of this study is to retrospectively evaluate treatment strategies for IBS used within primary Health care in Örebro Region.

DETAILED DESCRIPTION:
The defining features of IBS comprise the presence of recurrent abdominal pain in association with altered bowel habits (diarrhea, constipation or both), as stated in the Rome IV criteria. The spectrum, duration and severity of symptoms can range from inconvenient to incapacitating, and can prevent individuals from participating in everyday activities. Despite the prevalence of IBS, its management remains a challenge for global healthcare systems.

Treatment of IBS comprises, in summary, information to patients, dietary treatment, pharmacological treatment and psychological treatment. Pharmacological treatment includes antidepressants, bulking agents or fiber supplements, rifaximin, linaclotide, eluxadoline, loperamide, antispasmodics, prokinetics and probiotics.

Since the majority of patients with irritable bowel syndrome (IBS) are diagnosed and treated in primary care, the aim of this project is to investigate the adherence of general practitioners (GPs) to recommended therapeutic approaches for IBS.

In this study, data regarding therapeutic approaches will be collected retrospectively over the period of 2013-2019 by using the electronic patient register in Örebro Region. Patients will be identified by ICD-code K.58. The used treatments will be categorized in grade of recommendation as well as in strength of evidence. The efficacy of the used treatments will be evaluated, if possible. Over the counter agents, and lifestyle adjustments will not be evaluated.

The used treatments will be categorized in grade of recommendation (weak and strong) as well as in strength of evidence /very low, low, moderate and high). The eventual use of inappropriate treatments will be recorded as well. The efficacy of the used treatments will be, if possible, evaluated from the patient registers. The standardized and validated questionnaires IBS-Symptom Severity Score and IBS-Quality of Life scores are not routinely used within the primary health care. For this reason, the efficacy of the treatments will be categorized in "no effect, moderate effect and good effect".

Descriptive statistics will be used.

ELIGIBILITY:
Inclusion Criteria:

* All adult patients (both sexes) who were diagnosed with IBS according to ICD-10 in Region Örebro County 2013-2017.

Exclusion Criteria:

* Patients < 18 years or > 65 years.

Ages: 18 Years to 65 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with IBS within primary care of Region Örebro County 2013-2017.
Sampling Method: Non-Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 2021-11-29 (Estimated); Primary Completion 2023-05-31 (Estimated); Study Completion 2024-05-31 (Estimated)

PRIMARY OUTCOMES:
Adherence to guidelines of pharmacological treatment of IBS within primary care | 2013-2017
  The proportion of patients that have received pharmacological treatment according to guidelines for IBS within primary care.
Adherence to guidelines of non-pharmacological treatment of IBS within primary care | 2013-2017
  The proportion of patients that have received non-pharmacological treatment according to guidelines for IBS within primary care.

SECONDARY OUTCOMES:
Efficacy of treatment of IBS | 2013-2017
  Used treatments of IBS will be categorized in grade of recommendation as well as in strenght of evidence.
Use of inappropriate treatments of IBS | 2013-2017
  The prevalence of inappropriate treatment strategies of IBS within primary care will be recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Michiel van Nieuwenhoven, M.D. Ph.D., Principal Investigator — Region Örebro County

IPD SHARING:
Plan to Share IPD: Undecided